CLINICAL TRIAL: NCT03292406
Title: A Randomized, Double-blind, Multi-centre, Placebo-controlled, Parallel-arm Phase 2 Trial to Assess Safety, Efficacy and Pharmacokinetics of CD11301 0.03% and 0.06% Gel in the Treatment of Cutaneous T-Cell Lymphoma (CTCL), Stages IA, IB and IIA
Brief Title: A Safety, Efficacy and Pharmacokinetics Study of CD11301 for the Treatment of Cutaneous T-Cell Lymphoma (CTCL)
Acronym: CTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.03.SPR.104003
Record Dates: First submitted 2017-09-15; First posted 2017-09-25 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Cutaneous T Cell Lymphoma
Keywords: T-Cell; Lymphoma; Cutaneous; CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CD11301 Gel 0.06% (Experimental): Participants applied 0.06% CD11301 gel (up to 500 mg per dose) topically once daily, 3 to 5 times per week, for cycle 1 and 2 i.e. 24 weeks.
  Interventions: Drug: CD11301 0.06%
- CD11301 Gel 0.03% (Experimental): Participants applied 0.03% CD11301 gel (up to 500 mg per dose) topically once daily, 3 to 5 times per week, for cycle 1 and 2 i.e. 24 weeks.
  Interventions: Drug: CD11301 0.03%
- Placebo (Experimental): Participants applied placebo gel during cycle one followed by 0.03% CD11301 gel topically during cycle two once daily, 3 to 5 times per week, for 24 weeks.
  Interventions: Drug: Placebo; Drug: CD11301 0.03%

INTERVENTIONS:
Drug: Placebo — Non active ingredients of CD11301
  Arms: Placebo
Drug: CD11301 0.03% — Topical Gel
  Arms: CD11301 Gel 0.03%; Placebo
Drug: CD11301 0.06% — Topical Gel
  Arms: CD11301 Gel 0.06%

SUMMARY:
To assess the efficacy, safety and pharmacokinetics in participants treated with CD11301 gel vs. placebo for early stage CTCL (IA, IB, or IIA).

DETAILED DESCRIPTION:
To assess the efficacy and safety of two concentrations (0.03% and 0.06%) of CD11301 gel in the treatment of early stage CTCL (stage IA, IB, or IIA) versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of CTCL stage IA, IB, or IIA with biopsy within last 3 months
* Have BSA involvement corresponding to stages IA, IB or IIA CTCL with at least 3 distinct lesions

Exclusion Criteria:

* CTCL that is stage IIB or great or stage IIA with stage N2 with >5% circulating Sezary cells or CD8+ or large cell transformation or Progressive CTCL
* History of autoimmune disease
* Laboratory test values at screening outside of the normal range and judged clinically significant by the investigator
* Current participation in another clinical trial of a drug or device or past participation within 4 weeks before Baseline or participant is in exclusion period from a previous clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galderma R&D, Study Director — Galderma R&D
Locations (20):
- United States (10):
  - Galderma Investigational Site, Orange, California
  - Galderma Investigational Site, Palo Alto, California
  - Galderma Investigational Site, Farmington, Connecticut
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Boston, Massachusetts
  - Galderma Investigational Site, Durham, North Carolina
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Pittsburgh, Pennsylvania
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Houston, Texas
- France (3):
  - Galderma Investigational Site, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Galderma Investigational Site, Nantes, Pays de la Loire Region
  - Galderma Investigational Site, Paris, Île-de-France Region
- Germany (7):
  - Galderma Investigational Site, Mannheim, Baden-Wurttemberg
  - Galderma Investigational Site, Würzburg, Bavaria
  - Galderma Investigational Site, Krefeld, North Rhine-Westphalia
  - Galderma Investigational Site, Minden, North Rhine-Westphalia
  - Galderma Investigational Site, Münster, North Rhine-Westphalia
  - Galderma Investigational Site, Kiel, Schleswig-Holstein
  - Galderma Investigational Site, Berlin

IPD SHARING:
Plan to Share IPD: No
No intent to share information.

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 countries (France, Germany, USA) between 19 Dec 2017 to 17 Mar 2020. A total of 86 participants were randomized to 1 of the 3 treatment groups (placebo gel or CD11301 gel 0.03% or 0.06%) in a 1:1:1 ratio.
Pre-assignment Details: This study consisted of 2 cycles: Cycle 1 and Cycle 2. Each treatment cycle consisted of 8 weeks on treatment followed by 4 weeks without treatment. Cycle 1: drug product was applied on up to 5 percent (%) body surface area (BSA) and 10% BSA in cycle 2.
Period: Overall Study
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Started (Participants Randomized) | 30 | 28 | 28
Participants Treated | 30 | 28 | 27
Completed | 17 | 15 | 15
Not Completed | 13 | 13 | 13
Not completed — Progressive Disease | 6 | 3 | 4
Not completed — Adverse Event | 7 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 7 | 2
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo | Total
Number analyzed (Participants) | 30 | 28 | 28 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.43) | 56.8 (15.68) | 61.0 (14.21) | 59.5 (14.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 12 | 28
  Male | 22 | 20 | 16 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 29 | 27 | 26 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 28 | 27 | 24 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported Overall Response (Complete and Partial) of Target Treated Lesions Based on Modified Composite Assessment of Index Lesion Severity (mCAILS) Score at Week 12
Description: Overall response is defined as the number of participants that achieved a complete response (CR) or partial response (PR) as assessed by mCAILS. The mCAILS assessment total was derived from components collected on the case report form (CRF). Target treated lesions (1-5 lesions) were rated in erythema (0-8, where 0=no evidence and 8= very severe), scaling (0-8, where 0=no evidence and 8= very severe), plaque elevation (0-3, where 0=no evidence and 3= marked elevation), and size (scale=0-18, where 0= no measurable area and 18= size of lesion >300 centimeter [cm]^2). These 4 ratings were summed to create subtotals, 1 per lesion. The final mCAILS assessment score was the sum of these subtotals. Total summation Score: 0-50 where higher score indicated higher severity. Complete response is defined as a 100% decrease from baseline i.e. score of '0' on the mCAILS scale. Partial response is defined as at least a 50%, but less than 100%, decrease from baseline.
Time Frame: Week 12
Population: ITT Population included all randomized participants. Here, overall number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 4 | 7 | 1
Participants
  Complete Response | 0 | 2 | 0
  Partial Response | 4 | 5 | 1

2. Secondary Outcome: Number of Participants Reported Overall Response (OR) of Target Treated Lesions Based on Modified Severity-Weighted Assessment Tool (mSWAT) Score at Week 12
Description: OR is defined as the number of participants that achieved a complete response or partial response as assessed by mSWAT. mSWAT composite score involved the direct assessment of the BSA of each type of lesion (palm plus fingers of the participant= approximately 1% BSA) in each of 12 areas (Head, Neck, Anterior trunk, Arms, Forearms, Hands, Posterior trunk, Buttocks, Thighs, Legs, Feet, Groin) of the body, multiplying the sum of the BSA of each lesion type by a weighting factor (patch = 1, plaque = 2, and tumor = 3 or 4) and generating a sum of the subtotals of each lesion subtype. mSWAT score (0=no lesions; 400= lesions covering all areas). Complete response is defined as a 100% decrease from baseline. Partial response is defined as at least a 50%, but less than 100%, decrease from baseline, and with a tumor subscore of zero (no tumor).
Time Frame: Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 6 | 4 | 2
Participants
  Complete Response | 0 | 0 | 0
  Partial Response | 6 | 4 | 2

3. Secondary Outcome: Time to Participant's First Overall Response (Complete or Partial) of the Target Treated Lesions Based on the mCAILS Score
Description: Time to overall response (CR or PR) is the number of days from the start of drug application to the first documentation of objective response assessed by mCAILS Score. The 25th, 50th, and 75th percentiles were presented along with 95% confidence intervals using the log-log transformation. The mCAILS assessment total was derived from components collected on the case report form (CRF). Target treated lesions (1-5 lesions) were rated in erythema (0-8, where 0=no evidence and 8= very severe), scaling (0-8, where 0=no evidence and 8= very severe), plaque elevation (0-3, where 0=no evidence and 3= marked elevation), and size (scale=0-18, where 0= no measurable area and 18= size of lesion >300 centimeter [cm]^2). These 4 ratings were summed to create subtotals, 1 per lesion. The final mCAILS assessment score was the sum of these subtotals. Total summation Score: 0-50 where higher score indicated higher severity.
Time Frame: Up to Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 16 | 12 | 1
Days
  25th (95% CI) | 169 [84.0 to 169.0] | 85 [83.0 to 174.0] | NA [85.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.
  50th (95% CI) | 197 [169.0 to 257] | NA [169.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.
  75th (95% CI) | 257 [197.0 to 257] | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.

4. Secondary Outcome: Duration of Overall Response (Complete Response or Partial Response) Based on mCAILS Score
Description: The duration of overall response (complete or partial) of the target treated lesions based on the mCAILS score was calculated in days as: (date of first non-response after responding) - (date of response) + 1. The mCAILS assessment total was derived from components collected on the case report form (CRF). Target treated lesions (1-5 lesions) were rated in erythema (0-8, where 0=no evidence and 8= very severe), scaling (0-8, where 0=no evidence and 8= very severe), plaque elevation (0-3, where 0=no evidence and 3= marked elevation), and size (scale=0-18, where 0= no measurable area and 18= size of lesion >300 centimeter [cm]^2). These 4 ratings were summed to create subtotals, 1 per lesion. The final mCAILS assessment score was the sum of these subtotals. Total summation Score: 0-50 where higher score indicated higher severity.
Time Frame: Up to Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 12 | 10 | 1
Days
  25th (95% CI) | 133 [29.0 to 141.0] | NA [38.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.
  50th (95% CI) | 141 [133.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [38.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.
  75th (95% CI) | NA [133.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.

5. Secondary Outcome: Time to Progressive Disease Using mSWAT
Description: Progressive disease is defined as ≥ 25% increase in skin disease from baseline, or loss of response: in those with CR or PR, increase of skin score of greater than the sum of nadir plus 50% baseline score, Nadir is defined as the lowest skin score (best response).
Time Frame: Up to Week 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Days
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 26 | 21 | 24
Days
  25th (95% CI) | NA [170.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | 191 [85.0 to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | 93 [85.0 to 93.0]
  50th (95% CI) | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | 93 [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.
  75th (95% CI) | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | NA [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events. | 93 [NA to NA] — Missing quartiles and CIs were non-estimable due to a lack of events.

6. Secondary Outcome: Change From Baseline in Skindex-29 Survey Results at Week 12, 24 and 36
Description: Participants answered 30 questions as part of the Skindex-29 survey. A composite score and 3 sub scores were calculated from the results. Item 18 of the survey was not used in any scoring. First, answers to each item were given a numeric value: Never = 0; Rarely = 25; Sometimes = 50; Often = 75; All the time = 100. The items used to calculate each subscore were: Emotions: 3, 6, 9, 12, 13, 15, 21, 23, 26, and 28 (10 items), Symptoms: 1, 7, 10, 16, 19, 24, and 27 (7 items), Functioning: 2, 4, 5, 8, 11, 14, 17, 20, 22, 25, 29, and 30 (12 items). The composite score is the average of the 3 sub scores ranging from 0 (no effect)-100 (maximum effect), higher score corresponds to lower quality of life.
Time Frame: Week 12, 24 and Follow up (Week 36)
Population: ITT Population included all randomized participants. Here, overall number of participants analyzed signifies number of participants who were evaluable for this outcome measure and at specific category.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
Number analyzed (Participants) | 29 | 28 | 27
score on scale
  Week 12 | 1.93 (12.408) | -0.27 (8.583) | -1.58 (13.243)
  Week 24: number analyzed (Participants) | 23 | 26 | 24
  Week 24 | -2.16 (11.651) | -3.36 (9.816) | 0.58 (16.059)
  Week 36: number analyzed (Participants) | 22 | 19 | 20
  Week 36 | -3.30 (14.838) | -3.22 (8.340) | -0.34 (14.081)

ADVERSE EVENTS:
Time Frame: From start of the study drug administration up to end of the study (Week 72).
Description: Analysis was performed on safety population: randomized participants who applied the study medication at least once.
Arm/Group | CD11301 Gel 0.06% | CD11301 Gel 0.03% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 1/27
Serious Adverse Events (participants affected / at risk) | 2/30 | 2/28 | 1/27
Other Adverse Events (participants affected / at risk) | 30/30 | 28/28 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD11301 Gel 0.06% (N=30) | CD11301 Gel 0.03% (N=28) | Placebo (N=27)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD11301 Gel 0.06% (N=30) | CD11301 Gel 0.03% (N=28) | Placebo (N=27)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Bundle branch block left (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 1 (1) | 0 (0)
Application site erosion (General disorders) | 9 (19) | 3 (6) | 2 (3)
Application site ulcer (General disorders) | 8 (19) | 8 (13) | 2 (2)
Application site erythema (General disorders) | 7 (15) | 5 (6) | 2 (4)
Application site pain (General disorders) | 6 (8) | 3 (4) | 2 (2)
Influenza like illness (General disorders) | 6 (9) | 3 (4) | 2 (2)
Fatigue (General disorders) | 5 (7) | 5 (5) | 2 (2)
Application site pruritus (General disorders) | 4 (5) | 8 (12) | 4 (7)
Application site dermatitis (General disorders) | 4 (16) | 3 (9) | 1 (1)
Application site rash (General disorders) | 2 (4) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (5) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 3 (6)
Application site irritation (General disorders) | 1 (1) | 5 (15) | 1 (2)
Asthenia (General disorders) | 1 (1) | 2 (3) | 0 (0)
Application site eczema (General disorders) | 0 (0) | 0 (0) | 2 (3)
Application site inflammation (General disorders) | 0 (0) | 6 (16) | 1 (3)
Viral upper respiratory tract infection (Infections and infestations) | 4 (8) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (3) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (2) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (7) | 5 (6)
Headache (Nervous system disorders) | 7 (13) | 5 (8) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 5 (9) | 2 (8) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (10) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (6)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03292406/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT03292406/SAP_001.pdf